CLINICAL TRIAL: NCT07044427
Title: Investigation of Fall Risk Factors and Implementation of an Exercise Intervention for Prevention of Falls in Patients With Multiple Myeloma
Brief Title: Fall Risk Assessment and an Exercise Intervention for Prevention of Falls in Multiple Myeloma Patients
Acronym: Myfall
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Bethanien Krankenhaus gGmbH (Other)
Responsible Party: Principal Investigator, Ulrike Dapunt, Prof. Dr. med., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-045/2024
Record Dates: First submitted 2025-06-10; First posted 2025-07-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Fall Risk Factors; Strength Training Effects; Balance Training Effects
Keywords: Multiple Myeloma; Fall risk; pertubation training; strength training; Balance
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Other): Fall Prevention
  Interventions: Other: Strength and balance training in combination with a treadmill-based pertubation intervention

INTERVENTIONS:
Other: Strength and balance training in combination with a treadmill-based pertubation intervention — Patients receive a personalized home-based training plan with strength and balance exercises to be carried out three times a week for six months. In addition, treadmill-based pertubation training is carried out at 2 timepoints.

SUMMARY:
Approximately one third of the population over the age of 65 falls at least once a year. The risk of falling is in increased in older patients with tumor diseases. In addition to high treatment and care costs for the healthcare system, falls often lead to a decrease of quality of life, a reduction in physical performance and a loss of independence. Despite the high risk, falls in cancer patients have not yet been scientifically investigated in detail. For patients with multiple myeloma in particular, very little data is available on the prevalence, risk factors and effects of falls. In this study, a fall risk assessment is carried out in patients with multiple myeloma. Furthermore, a patient-specific training intervention for fall prevention will be implemented.

The aim of the study is to identify possible fall risk factors in multiple myeloma patients and to establish a structured exercise intervention that minimizes the risk of falls and injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma requiring therapy (at least 6 months of systemic therapy)
* ECOG status ≤ 3
* Age ≥18 years
* Patients who state that they want to carry out the training program at least 3 times/week and participate in the planned follow-up visits
* Ability to give informed consent
* Written consent to participate in the study
* Sufficient written and spoken German to complete the questionnaire

Exclusion Criteria:

* Any physical or mental limitations that would prevent participation in the training program or the planned follow-up checks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of at least 48 out of 72 training sessions with the focus on fall prevention within 24 weeks | From enrollement to the end of the training intervention at 6 months
  Patients will document the number of training sessions via an online training-app (Physiotec, Bad Wünnenberg, Germany). Feasibility is achieved if 48 of 72 possible training sessions were successfully completed.
Effectivity (fear of falling) | Evaluated at the beginning of the study and at the end of the study after 6 months
  Fear of falling will be evaluated by a validated questionnaire (FES-I, Falls Efficacy Scale-Inernational). The questionnaire contains 16 items scored on a four-point scale (1=not at all concerned to 4=very concerned). Scores >23 indicate high concern about falling.

CONTACTS AND LOCATIONS:
Overall Officials: Dapunt, Study Chair — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden Würtemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
* questionnaire results collected for each individual
  * functional test results collected for each individual

REFERENCES:
- [Background] Wildes TM, Fiala MA. Falls in older adults with multiple myeloma. Eur J Haematol. 2018 Mar;100(3):273-278. doi: 10.1111/ejh.13009. Epub 2018 Jan 8. PMID 29239009
- [Background] Wildes TM, Dua P, Fowler SA, Miller JP, Carpenter CR, Avidan MS, Stark S. Systematic review of falls in older adults with cancer. J Geriatr Oncol. 2015 Jan;6(1):70-83. doi: 10.1016/j.jgo.2014.10.003. Epub 2014 Oct 30. PMID 25454770
- [Background] Dapunt U, Ehret P, Paratte JL, Kuehl RM, Wiskemann J, Jager D, Muller-Tidow C, Raab MS, Goldschmidt H. A precision-based exercise program for patients with multiple myeloma. Eur J Haematol. 2023 Dec;111(6):930-937. doi: 10.1111/ejh.14106. Epub 2023 Sep 20. PMID 37727991
- [Background] Sattar S, Alibhai SM, Spoelstra SL, Fazelzad R, Puts MT. Falls in older adults with cancer: a systematic review of prevalence, injurious falls, and impact on cancer treatment. Support Care Cancer. 2016 Oct;24(10):4459-69. doi: 10.1007/s00520-016-3342-8. Epub 2016 Jul 22. PMID 27450557
- [Background] Pandya C, Magnuson A, Dale W, Lowenstein L, Fung C, Mohile SG. Association of falls with health-related quality of life (HRQOL) in older cancer survivors: A population based study. J Geriatr Oncol. 2016 May;7(3):201-10. doi: 10.1016/j.jgo.2016.01.007. Epub 2016 Feb 18. PMID 26907564